CLINICAL TRIAL: NCT03180645
Title: A Proof of Concept (POC) Clinical Study to Evaluate the Appearance of Fine Lines and Wrinkles on a Developmental Cosmetic Moisturising Cream in Healthy Subjects Presenting Visible Signs of Ageing
Brief Title: Proof of Concept Anti-ageing Clinical Study in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 207468
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Results first posted 2019-07-01 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-03

CONDITIONS: Skin Aging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test product/ No treatment (Other): Participants randomized to this arm will apply Test product at allocated sites and leave other sites untreated.
  Interventions: Other: Test product (Moisturising cream); Other: No treatment
- Test product/ Positive control (Other): Participants randomized to this arm will apply Test and positive product at allocated sites.
  Interventions: Other: Test product (Moisturising cream); Other: Positive control (Commercial market place moisturising cream)
- Positive control /No treatment (Other): Participants randomized to this arm will apply Positive product at allocated sites and leave other sites untreated.
  Interventions: Other: Positive control (Commercial market place moisturising cream); Other: No treatment

INTERVENTIONS:
Other: Test product (Moisturising cream) — Participants will be instructed to apply their assigned product to the randomly assigned side of the face, to include, the crow's feet area, cheek, forehead and chin twice daily (in the morning and evening).
  Arms: Test product/ No treatment; Test product/ Positive control
Other: Positive control (Commercial market place moisturising cream) — Participants will be instructed to apply their assigned product to the randomly assigned side of the face, to include, the crow's feet area, cheek, forehead and chin twice daily (in the morning and evening).
  Arms: Positive control /No treatment; Test product/ Positive control
Other: No treatment — No treatment
  Arms: Positive control /No treatment; Test product/ No treatment

SUMMARY:
The objective of this POC clinical study is to evaluate the moisturising effects on fine lines and wrinkles, texture, barrier function, hydration and elasticity delivered by 4 weeks of twice daily application of the test product on participants presenting visible signs of ageing.

DETAILED DESCRIPTION:
Participants who meet all the inclusion/exclusion criteria will be randomised to one of three treatment groups: test product/positive control, test product/no treatment or positive control/no treatment at the baseline visit. Product application within treatment group will be further randomised to either the right or left side of the face. Participants will apply one of the assigned treatments to one side of the face (left or right) and another assigned treatment to the other side of the face as per the randomisation schedule. Participants will be instructed to apply the assigned treatments twice daily (morning and evening, approximately 8-12 hours apart) for 4 weeks (28 days).

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form
* Good general and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant and relevant abnormalities in medical history or upon physical examination
* Females of childbearing potential who are, in the opinion of the investigator, practising a reliable method of contraception. Adequate contraception is defined as abstinence, oral contraceptive, either combined or progestogen alone OR injectable progestogen OR implants of levonorgestrel OR estrogenic vaginal ring OR percutaneous contraceptive patches OR intrauterine device or intrauterine system OR double barrier method (condom or occlusive cap [diaphragm or cervical vault caps] plus spermicidal agent [foam, gel, film, cream, suppository]) OR male partner sterilization prior to the female subject's entry into the study, and this male is the sole partner for that participant
* Willingness to actively participate in the study and to attend all scheduled visits
* Fitzpatrick phototype I-IV
* Visual Clinical Fitzpatrick Wrinkle Score 3- 6 in the eye (crow's feet) area on both sides of the face at screening and baseline
* Subjects with self-reported sensitive skin

Exclusion Criteria:

* Women who are known to be pregnant or who are intending to become pregnant over the duration of the study
* Women who are breast-feeding
* Any history of significant dermatological diseases or conditions or medical conditions known to alter skin appearance or physiologic response (e.g.diabetes,) which could, in the opinion of the Investigator, preclude topical application of the investigational products and/or interfere with the evaluations
* Change in contraception within the last 3 months
* Presence of open sores, pimples, cysts, irritated skin, hairs or tattoos at the application site
* Active dermatosis (local or disseminated) that might interfere with the results of the study
* Considered immune compromised
* Currently using any medication which in the opinion of the investigator, may affect the evaluation of the study product, or place the subject at undue risk
* Use of the following topical or systemic medications: immunosuppressants, antihistamines, non-hormonal anti-inflammatory drugs, and corticosteroids up to 2 weeks before screening visit
* Intention of using any oral or topical steroids
* Regular use of inhaled steroids (occasional use is permitted)
* Regular use of topical anti-itch medications (occasional use permitted; the product should be applied with an applicator but not to the proposed application areas
* Use of any topical drug or medication in the proposed application areas
* Intention of being vaccinated during the study period or has been vaccinated within 3 weeks of the screening visit
* Currently receiving allergy injections, or received an allergy injection within 7 days prior to Visit 1, or expects to begin injections during study participation
* Blepharitis, conjunctivitis, uveitis
* Topical ocular treatment within the last month
* Aesthetic, cosmetic or dermatological treatment on the face within the last 3 months
* Intense sun exposure, Ultra Violet-treatments or tanning salon visit within the last 2 weeks
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 14 days of the screening visit
* Previous participation in this study
* Recent history (within the last 5 years) of alcohol or other substance abuse
* An employee of the sponsor or the study site or members of their immediate family
* A smoker

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 72 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-04-21 (Actual); Study Completion 2017-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Schenefeld, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nisbet S, Mahalingam H, Gfeller CF, Biggs E, Lucas S, Thompson M, Cargill MR, Moore D, Bielfeldt S. Cosmetic benefit of a biomimetic lamellar cream formulation on barrier function or the appearance of fine lines and wrinkles in randomized proof-of-concept clinical studies. Int J Cosmet Sci. 2019 Feb;41(1):1-11. doi: 10.1111/ics.12499. Epub 2019 Feb 22. PMID 30414275

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All the participants were enrolled at one center in Germany.
Pre-assignment Details: A total of 86 participants were screened, out of which 14 did not meet study criteria, remaining 72 participants were randomized to the study.
Groups:
- Test Product/ No Treatment: Participants randomized to this arm applied Test product at allocated side and left other side untreated.
- Test Product/ Positive Control: Participants randomized to this arm applied Test and positive product at allocated sides.
- Positive Control /No Treatment: Participants randomized to this arm applied Positive product at allocated side and left other side untreated.
Period: Overall Study
Arm/Group | Test Product/ No Treatment | Test Product/ Positive Control | Positive Control /No Treatment
Started | 24 | 24 | 24
Completed | 24 | 23 | 22
Not Completed | 0 | 1 | 2
Not completed — Adverse Event | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Safety population (N=72), included all participants who applied any of the study products.
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Product/ No Treatment | Test Product/ Positive Control | Positive Control /No Treatment | Total
Number analyzed (Participants) | 24 | 24 | 24 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 24 | 24 | 72
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 24 | 72
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 24 | 24 | 24 | 72
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Ra (a dermaTOP Parameter), of Test Product Treated Versus (vs.) Untreated Side at Day 29
Description: Using fringe projection and optical triangulation techniques, the 3D (three dimensional) surface structure of a designated investigational skin site on each side of the face was captured as an in vivo measurement using dermaTOP. From the captured 3D structure, roughness parameters were calculated. Ra is usually used for wrinkle assessments, representing the finer skin structure (Ra). Ra was the average deviation of the profile from the mean line (arithmetic mean of the absolute values of the point's heights).
Time Frame: At Baseline and Day 29
Population: Analysis population was ITT (N=70) population included all participants who were randomized into the study and had at least one post-baseline clinical assessment available.
Measure: Mean (Standard Deviation); unit: Micro meter (µm)
Groups:
- Test Product: Data of this arm included all allotted sides of the face of the participants where test product was applied during the study.
- No Treatment: Data of this arm Included all allotted sides of the face of the participants which were left untreated during the study.
Arm/Group | Test Product | No Treatment
Number analyzed (Participants) | 47 | 46
Micro meter (µm) | -1.90 (4.245) | -0.12 (3.478)
Statistical Analysis 1: Comparison: Test Product vs No Treatment; Test type: Other; p = 0.0638, ANCOVA; Analysis model (ANCOVA) included participant as random effect, treatment arm and side of the face as fixed effects and baseline value as covariate; Least square (LS) mean difference = -1.07, 95% CI 2-sided [-2.21 to 0.06] — Difference is the first named treatment adjusted (LS) mean change from baseline minus the second named treatment adjusted mean change from baseline

2. Secondary Outcome: Change From Baseline in Ra (a dermaTOP Parameter), of Test Product Treated vs. Untreated Side at Day 15
Description: Using fringe projection and optical triangulation techniques, the 3D surface structure of a designated investigational skin site on each side of the face was captured as an in vivo measurement using dermaTOP. From the captured 3D structure, roughness parameters were calculated. Ra is usually used for wrinkle assessments, representing the finer skin structure (Ra). Ra was the average deviation of the profile from the mean line (arithmetic mean of the absolute values of the point's heights).
Time Frame: At Baseline and Day 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Test Product | No Treatment
Number analyzed (Participants) | 48 | 46
µm | -0.65 (4.487) | -0.18 (3.237)

3. Secondary Outcome: Change From Baseline in Ra (a dermaTOP Parameter), of Positive Control Treated vs. Untreated Side at Day 15 and 29
Description: Using fringe projection and optical triangulation techniques, the 3D surface structure of a designated investigational skin site on each side of the face was captured as an in vivo measurement using dermaTOP. From the captured 3D structure, roughness parameters were calculated. Ra is usually used for wrinkle assessments, representing the finer skin structure (Ra). Ra is the average deviation of the profile from the mean line (arithmetic mean of the absolute values of the point's heights).
Time Frame: At Baseline, Day 15 and 29
Population: Analysis population was ITT (N=70) population included all participants who were randomized into the study and had at least one post-baseline clinical assessment available. Here, number analyzed signifies number of participants who were evaluable at the specified time points.
Measure: Mean (Standard Deviation); unit: µm
Groups:
- Positive Control: Data of this arm Included all allotted sides of the face of the participants where positive control was applied during the study.
Arm/Group | Positive Control | No Treatment
Number analyzed (Participants) | 46 | 46
µm
  Day 15 | 0.18 (2.543) | -0.18 (3.237)
  Day 29: number analyzed (Participants) | 45 | 46
  Day 29 | -0.13 (3.461) | -0.12 (3.478)

4. Secondary Outcome: Change From Baseline in Rz (a dermaTOP Parameter) at Day 15 and 29
Description: Using fringe projection and optical triangulation techniques, the 3D surface structure of a designated investigational skin site on each side of the face was captured as an in vivo measurement using dermaTOP. From the captured 3D structure, roughness parameters were calculated. Rz usually used for wrinkle assessments, representing the rough structure, such as wrinkles. Rz was an average of the 5 sub-profiles (peak to valley heights) local maximum. From each local profile the peak to peak height value is calculated; the average of the 5 peak to peak height values was Rz.
Time Frame: At Baseline, Day 15 and 29
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Test Product | Positive Control | No Treatment
Number analyzed (Participants) | 48 | 46 | 46
µm
  Day 15 | -1.92 (18.864) | 0.97 (10.508) | -1.46 (13.194)
  Day 29: number analyzed (Participants) | 47 | 45 | 46
  Day 29 | -7.01 (18.395) | -0.55 (14.144) | -1.08 (15.279)

5. Secondary Outcome: Change From Baseline in Sa (dermaTOP Parameters) at Day 15 and 29
Description: Using fringe projection and optical triangulation techniques, the 3D surface structure of a designated investigational skin site on each side of the face was captured as an in vivo measurement using dermaTOP. The 3D skin surface profile was calculated from the position of the fringes in combination with the Gray values of each pixel. From the captured 3D structure, roughness parameters were calculated. Sa was the arithmetic average of the absolute (non- signed) heights of the topography points. Sa was the 3D Area -Equivalent of 2D profile roughness parameter Ra.
Time Frame: At Baseline, Day 15 and 29
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Test Product | Positive Control | No Treatment
Number analyzed (Participants) | 48 | 46 | 46
µm
  Day15 | -0.60 (4.426) | 0.17 (2.646) | -0.08 (3.291)
  Day 29: number analyzed (Participants) | 47 | 45 | 46
  Day 29 | -1.83 (4.076) | -0.21 (3.354) | -0.26 (3.433)

6. Secondary Outcome: Change From Baseline in Stm (dermaTOP Parameters), at Day 15 and 29
Description: Using fringe projection and optical triangulation techniques, the 3D surface structure of a designated investigational skin site on each side of the face was captured as an in vivo measurement using dermaTOP. The 3D skin surface profile was calculated from the position of the fringes in combination with the Gray values of each pixel. From the captured 3D structure, roughness parameters were calculated. Stm was an average of the 5x5 sub-areas (peak to valley heights) local maximum: The surface was virtually divided into 25 sub-surfaces (5 rows, 5 columns); from each local surface the peak to peak height value is calculated; the average of the 25 peak to height values was Stm.
Time Frame: At Baseline, Day 15 and 29
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Test Product | Positive Control | No Treatment
Number analyzed (Participants) | 48 | 46 | 46
µm
  Day 15 | 5.81 (62.571) | 5.35 (29.232) | -2.02 (33.670)
  Day 29: number analyzed (Participants) | 47 | 45 | 46
  Day 29 | -12.89 (47.901) | 0.23 (35.323) | -3.27 (35.025)

7. Secondary Outcome: Change From Baseline in Clinical Fitzpatrick Wrinkle Score, at Day 15 and 29
Description: A blinded, trained and qualified examiner performed Clinical Fitzpatrick Wrinkle Score assessments by visually grading the crow's feet area under standard conditions of illumination. Fitzpatrick Wrinkle Scores range between 1-9 where 1-3= Fine wrinkles, 4-6= Fine to moderate depth wrinkles, a moderate number of wrinkles, 7-9= Fine to deep wrinkles, numerous lines, with or without redundant skin folds. Low value indicated better results.
Time Frame: At Baseline, Day 15 and 29
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Test Product | Positive Control | No Treatment
Number analyzed (Participants) | 48 | 46 | 46
Score on a scale
  Day 15 | -0.33 (0.559) | -0.28 (0.544) | -0.15 (0.420)
  Day 29: number analyzed (Participants) | 47 | 45 | 46
  Day 29 | -0.51 (0.688) | -0.58 (0.583) | -0.22 (0.664)

8. Secondary Outcome: Change From Baseline in Instrumental Corneometer Values, at Day 15 and 29
Description: Measurement of Stratum Corneum (SC) hydration was performed by the electrical capacitance method with a Corneometer. The measuring principle was based on changes in the capacitance of the measuring head, functioning as a condensator. An electric field was created between gold conductors to enable the dielectricity of the SC to be measured. Because the dielectricity varies as a function of the skin's water content, the SC moisturisation was measured. Higher value of corneometery indicates high moisture content.
Time Frame: At Baseline, Day 15 and 29
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Instrumental units (I.U)
Arm/Group | Test Product | Positive Control | No Treatment
Number analyzed (Participants) | 48 | 46 | 46
Instrumental units (I.U)
  Day 15 | 6.12 (7.566) | 7.13 (8.238) | -1.09 (10.813)
  Day 29: number analyzed (Participants) | 47 | 45 | 46
  Day 29 | 8.30 (8.865) | 10.03 (10.070) | 1.62 (10.186)

9. Secondary Outcome: Percent Improvement From Baseline in Skin Texture Rankings Based on Lay Grader Assessment of High Resolution Images at Day 29
Description: High resolution images of the left and right side of each participant's whole half-face were taken at baseline and Day 29. Each blinded image pair was randomly displayed on a color-calibrated screen and assessed by a panel of lay graders, who ranked each image based on texture, defined as pores, smoothness and unevenness, on a scale of: 1 = better; or 2 = worse (lower score indicated improvement). The total proportion of improvement (from all lay graders) on Day 29 than baseline is reported for this endpoint.
Time Frame: At Baseline and Day 29
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percent of improvement ratings
Groups:
- Negative Control: Data of this arm Included all allotted sides of the face of the participants which were left untreated during the study.
Arm/Group | Test Product | Positive Control | Negative Control
Number analyzed (Participants) | 47 | 45 | 46
Percent of improvement ratings | 41.49 [38.60 to 44.43] | 39.54 [36.61 to 42.52] | 40.58 [37.67 to 43.54]

10. Secondary Outcome: Change From Baseline in Instrumental Cutometer Parameters R5, at Day 15 and 29
Description: The Cutometer measures elasticity of the upper skin layer using negative pressure which deforms the skin mechanically. Negative pressure was created in the device and the skin was drawn into the aperture of the probe and after a defined time released again. Inside the probe, the penetration depth was determined by a non-contact optical measuring system. The light intensity varies due to the penetration depth of the skin. The resistance of the skin to the negative pressure (firmness) and its ability to return into its original position (elasticity) was displayed as curves (penetration depth in mm/time) in real time during the measurement. This measurement principle provides information about the elastic and mechanical properties of the skin surface and enables objective quantification of skin ageing. R5 (net elasticity): the elastic portion of the suction part versus the elastic portion of the relaxation part.
Time Frame: At Baseline, Day 15 and 29
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Ratio (unitless)
Arm/Group | Test Product | Positive Control | No Treatment
Number analyzed (Participants) | 48 | 46 | 46
Ratio (unitless)
  Day 15 | 0.05 (0.132) | 0.01 (0.121) | -0.05 (0.104)
  Day 29: number analyzed (Participants) | 47 | 45 | 46
  Day 29 | 0.08 (0.144) | 0.05 (0.139) | 0.03 (0.113)

11. Secondary Outcome: Change From Baseline in Instrumental Cutometer Parameter R7, at Day 15 and 29
Description: The Cutometer measures elasticity of the upper skin layer using negative pressure which deforms the skin mechanically. Negative pressure was created in the device and the skin was drawn into the aperture of the probe and after a defined time released again. Inside the probe, the penetration depth was determined by a non-contact optical measuring system. The light intensity varies due to the penetration depth of the skin. The resistance of the skin to the negative pressure (firmness) and its ability to return into its original position (elasticity) are displayed as curves (penetration depth in mm/time) in real time during the measurement. This measurement principle provides information about the elastic and mechanical properties of the skin surface and enables objective quantification of skin ageing. R7: Portion of the elasticity compared to the complete curve values.
Time Frame: At Baseline, Day 15 and 29
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Ratio (unitless)
Arm/Group | Test Product | Positive Control | No Treatment
Number analyzed (Participants) | 48 | 46 | 46
Ratio (unitless)
  Day 15 | 0.02 (0.079) | 0.01 (0.075) | -0.03 (0.063)
  Day 29: number analyzed (Participants) | 47 | 45 | 46
  Day 29 | 0.03 (0.093) | 0.02 (0.079) | 0.02 (0.067)

12. Secondary Outcome: Change From Baseline in Trans-Epidermal Water Loss (TEWL) at Day 15 and 29
Description: TEWL measuring principle was based on water vapour gradient determination between two pairs of sensors (temperature and relative humidity) placed at different distances perpendicularly to the skin. Measurements were taken in triplicate and then an average (mean) reading was calculated on the left and right Sub-ocular/ Cheek Area directly from the corner of the eyes onto the middle of the cheekbone. A decrease in TEWL corresponds to an improved skin barrier function.
Time Frame: At Baseline, Day 15 and 29
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: gram (g)/meter^2 (m)/hour
Arm/Group | Test Product | Positive Control | No Treatment
Number analyzed (Participants) | 48 | 46 | 46
gram (g)/meter^2 (m)/hour
  Day 15 | -4.17 (4.904) | -5.98 (4.994) | -2.02 (4.713)
  Day 29: number analyzed (Participants) | 47 | 45 | 46
  Day 29 | -5.18 (3.719) | -6.62 (5.791) | -3.00 (4.564)

ADVERSE EVENTS:
Time Frame: Approximately 30 days
Description: All treatment emergent adverse events (AEs) were reported in this section. Skin-related AEs counted under one or both treatment groups that the subject received based on the application site(s). Non-skin related adverse events counted under both treatment groups that the subject received. Each adverse event was counted only once in the Overall column irrespective of whether it was skin related or not.
Groups:
- Overall Participants: All randomized participants were included in the baseline assessment and received test product (moisturizing cream), positive control and no treatment.
Arm/Group | Test Product | Positive Control | No Treatment | Overall Participants
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48 | 0/48 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48 | 0/48 | 0/72
Other Adverse Events (participants affected / at risk) | 12/48 | 10/48 | 11/48 | 17/72
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Test Product (N=48) | Positive Control (N=48) | No Treatment (N=48) | Overall Participants (N=72)
Headache (Nervous system disorders) | 6 | 4 | 4 | 7
BURNING SENSATION (Nervous system disorders) | 0 | 2 | 0 | 2
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 2
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 2
SKIN TIGHTNESS (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 1 | 0 | 1 | 1
OTITIS MEDIA (Infections and infestations) | 1 | 0 | 1 | 1
ORAL HERPES (Infections and infestations) | 0 | 1 | 1 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
DRY EYE (Eye disorders) | 1 | 0 | 1 | 1
SLEEP DISORDER (Psychiatric disorders) | 1 | 0 | 1 | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
SCRATCH (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-03-24): https://cdn.clinicaltrials.gov/large-docs/45/NCT03180645/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-12): https://cdn.clinicaltrials.gov/large-docs/45/NCT03180645/SAP_001.pdf